CLINICAL TRIAL: NCT05295251
Title: The Commonest Medical, Surgical, and Oncological Causes of Acute Abdomen in Adults With COVID-19. A Prospective Observational Study.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: acute abdomen in covid
Record Dates: First submitted 2022-03-24; First posted 2022-03-25 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Acute Abdomen
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medical ,oncological and surgical treatment of cases of acute abdomen — medical treatment and surgical intervention during covid-19 pandemic

SUMMARY:
Coronaviruses are a large family of viruses that can cause mild to severe respiratory infections. 2019-nCoV is a novel coronavirus that was discovered in Wuhan, China. Since its discovery in humans in late 2019, it has had a global, rapid spread. Dry cough, fever, and fatigue are the most common symptoms in the first two to 14 days after exposure.

At the moment, it is unknown how common gastrointestinal symptoms are. However, COVID-19's initial clinical presentations have become more evident as the pandemic has progressed and case data has been gathered, and literature suggests that digestive symptoms are prevalent .

In a recent systematic review and meta-analysis of 47 studies involving 10,890 patients with COVID-19, the pooled prevalence of gastrointestinal symptoms were 7.7 % for diarrhea, 7.8% for nausea/vomiting, and 2.7% for abdominal pain. Only a few cases of isolated abdominal pain have been reported.

A wide range of diseases can cause acute abdominal pain, and diagnosing them can be difficult. The examining physician should prioritize life-threatening conditions that may necessitate immediate surgical intervention with such a broad differential diagnosis to avoid further mortality or morbidity. The objective of this study was to determine the characteristics, incidence, severity and of acute abdominal pain (medical and surgical causes) during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Coronaviruses are a large family of viruses that can cause mild to severe respiratory infections. 2019-nCoV is a novel coronavirus that was discovered in Wuhan, China. Since its discovery in humans in late 2019, it has had a global, rapid spread. Dry cough, fever, and fatigue are the most common symptoms in the first two to 14 days after exposure.

At the moment, it is unknown how common gastrointestinal symptoms are. However, COVID-19's initial clinical presentations have become more evident as the pandemic has progressed and case data has been gathered, and literature suggests that digestive symptoms are prevalent .

In a recent systematic review and meta-analysis of 47 studies involving 10,890 patients with COVID-19, the pooled prevalence of gastrointestinal symptoms were 7.7 % for diarrhea, 7.8% for nausea/vomiting, and 2.7% for abdominal pain. Only a few cases of isolated abdominal pain have been reported.

A wide range of diseases can cause acute abdominal pain, and diagnosing them can be difficult. The examining physician should prioritize life-threatening conditions that may necessitate immediate surgical intervention with such a broad differential diagnosis to avoid further mortality or morbidity. The objective of this study was to determine the characteristics, incidence, severity and of acute abdominal pain (medical and surgical causes) during the COVID-19 pandemic.

Acute abdominal pain in COVID-19 patients poses a diagnostic quandary for clinicians. Delays in treating an acute abdomen can lead to severe complications and even death. In contrast, performing unnecessary surgery on COVID-19 patients results in increased morbidity and mortality, increased strain on healthcare resources, and an increased risk of exposure for healthcare workers in operative fields. This study aimed to determine the characteristics, incidence and severity, and of various medical and surgical causes of acute abdomen in COVID-19. According to our study, gastritis is the most common medical cause of acute abdomen (19.2%). While acute appendicitis (42.4%), acute cholecystitis (11%), and biliary colic (9.8%) are the most frequently encountered surgical causes of acute abdomen, acute pancreatitis occurred in (3%) of cases and mainly was benign in course. Except for acute appendicitis, intestinal ischemia and liver abscesses, the severity of all causes of acute abdomen did not worsen.

Abdominal pain is a less frequent symptom of COVID-19 infection than anorexia, nausea/vomiting, or diarrhea. Abdominal pain is prevalent in 3.9-6.8% of the population .

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* male and female
* covid-19 positive
* acute abdomen

Exclusion Criteria:

* < 18 years
* unsure diagnosis of covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients > 18 years of age, both sexes, admitted to the emergency department or already admitted but complaining of an acute abdomen, and diagnosed with COVID-19 using a thoracic computed tomography (CT) scan and/or reverse transcription polymerase chain reaction (RT-PCR) of SARS-CoV-2 RNA, as per the Institute Pasteur protocol and WHO technical guidelines [8]. Patients younger than 18 years of age and those who were not confirmed to be COVID-19 positive were excluded from the study. All patients who underwent chest computed tomography (CT) and a comprehensive panel of routine laboratory tests, which included a complete blood count, urinalysis, blood biochemistry, and blood coagulation function.
Sampling Method: Probability Sample
Enrollment: 910 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
characteristic, severity and incidence of acute abdomen | 2 years
  incidence in %

CONTACTS AND LOCATIONS:
Overall Officials: Alnaimy A alnaimy, Phd, Principal Investigator — Zagazig University
Locations (1):
- Tamer Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided